CLINICAL TRIAL: NCT00348738
Title: The Influence of the Pre-Therapeutic Increase in the Hemoglobin Level in the Blood Through Erythropoietin to the Therapy Results of the Primary Radiation Therapy for Carcinoma of the Cervix
Brief Title: Impact of Erythropoietin Administration During Definitive Cervix Cancer Radiotherapy on Treatment Outcome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OEGRO54
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Cervix Cancer
Keywords: radiotherapy; clinical trial; erythropoietin; cervix cancer; Phase III; 2 Arms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients assigned to this group are receiving Erythropoietin medication
  Interventions: Drug: Erythropoietin
- 2 (No Intervention): control group receiving no treatment

INTERVENTIONS:
Drug: Erythropoietin — Administration of 10.000 I.U Erythropoeitin SQ 3x/week, two weeks prior to radiation therapy until a haemoglobin concentration of >14g/dl, <15g/dl is reached or until the end of the radiation therapy.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether an increase of blood haemoglobin levels through the substitution of erythropoietin during radiotherapy treatment of cervix cancer patients results in improvement for disease specific survival, tumor response and local control.

DETAILED DESCRIPTION:
Definitive radiotherapy is the treatment of choice for patients with locally advanced cervix cancer. Low pre-therapeutic values of the intratumoral pO2 are associated with significantly worse therapeutic outcome and the blood hemoglobin levels correlate positively with the intratumoral pO2. Successful augmentation of hemoglobin levels by way of transfusion leads to improvement of therapeutic results. Therefore, a pre-therapeutic transfusion therapy is carried out routinely at a number of hospitals; however this therapy is due to its cost and risks limited to patients with an initial hemoglobin level of < 10 g/dl. To avoid transfusions and to increase patients wellbeing, the efficacy and tolerability of erythropoietin was tested, when administered to increase the lowered hemoglobin levels in tumor patients. The question is, whether or not it is possible, to regularly raise the blood hemoglobin levels in patients with carcinoma of the cervix by administering erythropoietin. If a normal (>12 g/dl) or rather an upper-normal (>14 g/dl) hemoglobin level is reached, then the tumor oxygenation and thus also the response to radiation could be positively influenced. The objective of this study is to improve the response and control rates as well as the disease free survival rates in female patients with primary carcinoma of the cervix within the scope of the curative radiation therapy. The test hypothesis is that by administering erythropoietin the hemoglobin levels are increased and through this increase the response of the tumor to radiation therapy will be improved.

Comparison(s): A prospective, randomized, multi-centric group of female patients treated with Erythropoietin is compared to a parallel stratified control group receiving no treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven cervix cancer (FIGO stage I-IVA)
* Age of 19-80 years
* initial blood level of hemoglobin <= 14 g/dl
* patients who gave their informed consent

Exclusion Criteria:

* Karnofsky-Index < 50 %
* known intolerance of erythropoietin
* FIGO stage IVB
* blood transfusion within the last four weeks
* neoadjuvant chemotherapy
* previous radiation therapy of the abdomen

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2000-07; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
remission rate 3 months after completion of the radiation therapy | 3 months
local control rate | 2 years
Disease specific survival | 2 years

SECONDARY OUTCOMES:
The extent of increase in hemoglobin levels during the treatment with erythropoietin. | Duration of treatment
The need of transfusion during the treatment. | Duration of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Poetter, Prof., M.D., Study Chair — Department of Radiotherapy and Radiobiology-Medical University of Vienna
Locations (4):
- Austria (4):
  - Department of Radiotherapy-University Hospital of Innsbruck, Innsbruck
  - Department of Radiotherapy-University Hospital of Salzburg, Salzburg
  - Department of Radiotherapy and Radiobiology-Medical University of Vienna, Vienna
  - Department of Radiotherapy-Hospital of Hietzing, Vienna

REFERENCES:
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Sobel E, Rose GS, Thomas G, Carlson JW. Association of hemoglobin level with survival in cervical carcinoma patients treated with concurrent cisplatin and radiotherapy: a Gynecologic Oncology Group Study. Gynecol Oncol. 2004 Aug;94(2):495-501. doi: 10.1016/j.ygyno.2004.04.008. PMID 15297194
- [Background] Vaupel P, Thews O, Mayer A, Hockel S, Hockel M. Oxygenation status of gynecologic tumors: what is the optimal hemoglobin level? Strahlenther Onkol. 2002 Dec;178(12):727-31. doi: 10.1007/s00066-002-1081-x. PMID 12491062
- [Background] Knocke TH, Weitmann HD, Feldmann HJ, Selzer E, Potter R. Intratumoral pO2-measurements as predictive assay in the treatment of carcinoma of the uterine cervix. Radiother Oncol. 1999 Nov;53(2):99-104. doi: 10.1016/s0167-8140(99)00139-5. PMID 10665785